CLINICAL TRIAL: NCT04582747
Title: Urinary Biomarkers for the Prediction of Acute Kidney Injury Following Major Abdominal Surgery
Brief Title: Acute Kidney Injury - Biomarkers in Major Abdominal Surgery
Acronym: AKI-BioMAS
Status: Completed | Type: Observational
Sponsor: Royal Surrey County Hospital NHS Foundation Trust (Other)
Responsible Party: Sponsor
Other Study IDs: AKI-BioMAS
Record Dates: First submitted 2019-09-18; First posted 2020-10-12 (Actual); Last update posted 2020-10-12 (Actual); Status verified 2020-10

CONDITIONS: Acute Kidney Injury
MeSH Terms: conditions — Acute Kidney Injury

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Urine samples from post-operative abdominal surgery patients
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Major abdominal Surgery patients: Major Abdominal Surgery Patients
  Interventions: Diagnostic Test: Urinary Biomarkers (NGAL, DKK-3, IGFBP-7/TIMP-2, KIM-1)

INTERVENTIONS:
Diagnostic Test: Urinary Biomarkers (NGAL, DKK-3, IGFBP-7/TIMP-2, KIM-1) — Validation of Urinary biomarker tests for the rapid prediction of AKI.
  No intervention is being proposed as part of the study. Concentrations of Urinary biomarkers will be obtained post operatively. These concentrations will be assessed to ascertain their predictive ability for the development of Acute Kidney Injury post-operatively.

SUMMARY:
To validate Urinary Biomarkers for the prediction of AKI in major abdominal surgery patients

DETAILED DESCRIPTION:
Background

Surgery is a risk factor for acute kidney Injury (AKI). Surgery exposes patients to hypotension, sepsis, the infusion of blood products, ischaemia, oxidative stress and reperfusion injury.

Patients who develop AKI post operatively are susceptible to fluid overload, infections, and cardiac events. AKI confers an increased risk of chronic kidney disease and mortality. Studies assessing rates of AKI in general surgical patients place the frequency at 1-14%.

Established methods of assessing for AKI - products of nitrogen breakdown and urine output - have limitations. Serum creatinine and urea are affected by sex, nutritional status, blood in the gastrointestinal tract, and fluid resuscitation. Rises in serum creatinine become apparent once glomerular filtration has reduced by half. This potentially delays the use of reno-protective strategies.

Novel biomarkers have been investigated. These aim to verify the use of renal biomarkers as a method of identifying AKI more rapidly: It is hoped that reno-protective strategies could be adopted sooner.

Much work has concerned cardiac and transplant surgery. AKI rates have been quoted as high as 30% in this cohort. Results were initially encouraging for various biomarkers. One biomarker (Insulin like growth factor binding protein number 7 / Tissue inhibitor of metalloproteinases 2 - IGFBP-7/TIMP-2) has therefore been incorporated into Enhanced Recovery Programmes in such patients.

While research in cardiac and transplant surgery has been extensive, it has been limited with regards to abdominal surgery. Although rates of AKI are lower in this cohort, they still bear a significant burden of disease. At present, no biomarker has been found to be clinically useful in this setting.

Study Objectives

Primary

The validation of Urinary Biomarkers for use in the prediction of AKI in major abdominal surgery patients

Secondary

To assess the role different surgical sub-types and peri-operative factors have in causing AKI in Major Abdominal Surgery patients

Trial design

This is an observational study that will assess the use of Urinary biomarkers against conventional methods of assessing for AKI, the Kidney Disease, Improving Global Outcomes (KDIGO) criteria. The KDIGO criteria is based on increases in serum creatinine and reduction in urine output.

The biomarkers are:

IGFBP-7/TIMP-2 Neutrophil Gelatinase Associated Lipocalin (NGAL) Kidney Injury Molecule 1 (KIM-1) Dickkopf related protein 3 (DKK-3)

All patients undergoing major elective general surgery, and major abdominal gynaecological surgery will be included. All patients will have a urine sample taken 4 hours post operatively. This sample will be tested using the biomarkers. Written consent will be obtained from all participants.

The consent form has been designed with help of 10 surgical inpatients and 4 surgical nurses to ensure ease of understanding and a lack of medical jargon.

No changes are required to standard patient care. The urine sample obtained will be a catheter specimen.

Comparison of the novel biomarkers against conventional methods will be conducted using the KDIGO criteria. This entails regular urine output measurement, assessment of blood urea, electrolytes, and estimated glomerular filtration rate. Data regarding patient, operative and post-operative characteristics will be recorded on a purpose-built secure hospital intranet database.

Data Analysis

Performance of the biomarkers will be assessed using multiple logistic regression, and by conducting 'area under the receiver-operator curve (AUROC)' analysis. A risk prediction model will be created based on patient factors strongly associated with the primary endpoint. The performance of the risk prediction model will be assessed as a standalone test and in conjunction with the novel biomarker tests.

The sample size was calculated on the basis of previously published AUROC values for the test, the expected prevalence of AKI, and a desire for a 95% confidence interval around the calculated AUROC estimate for the study. This results in a target sample size of 471.

Hoped Aims of Research

The researchers hope that a novel test is found that can identify AKI sooner in an at-risk cohort of patients. If so, a further trial is intended: post-operative patients who are positive to the novel test will be randomised to a kidney protective 'bundle', and rates of AKI compared.

Ultimately, the intention is to greatly reduce a significant cause of post-operative morbidity, surgical complications, and mortality, through the judicious use of a non-invasive test.

ELIGIBILITY:
Inclusion Criteria:

* • Patients aged over 18 undergoing major Hepatobiliary, Oesophagogastric, Colorectal or abdominal Gynaecological Surgery at the Royal Surrey County Hospital. Patients undergoing Liver Transplant Surgery at King's College Hospital

  * Be able to provide informed consent

Exclusion Criteria:

* Patients requiring renal replacement therapy prior to the study
* Patients with pre-operative AKI
* Patients without baseline creatinine measurements
* Day case surgery
* Patients unable to consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients undergoing major elective general surgery, and major abdominal gynaecological surgery will be included
Sampling Method: Non-Probability Sample
Enrollment: 500 (Actual)
Dates: Start 2018-07-03 (Actual); Primary Completion 2020-03-03 (Actual); Study Completion 2020-03-03 (Actual)

PRIMARY OUTCOMES:
The diagnostic performance (expressed as the 'Area under the receiver-operator curve') of Urinary Biomarkers for the rapid prediction of Acute Kidney Injury in Major Abdominal Surgery patients. | The study aims to assess the diagnostic performance of the biomarkers to predict the development of AKI within 3 days of the surgical procedure. Renal function will be assessed daily within this time frame.
  Conventional renal function measurement - assessing blood creatinine - often does not identify Acute Kidney Injury until 48 hours has passed from the time of insult.
  It is hypothesised that the studied urinary biomarkers may be able to identify patients who develop AKI 4 hours post-operatively.

CONTACTS AND LOCATIONS:
Locations (1):
- Royal Surrey County Hospital, Guildford, Surrey, United Kingdom

IPD SHARING:
Plan to Share IPD: No
Participants are anonymised in the study. Demographic and clinical data will be provided as part of the study write up